CLINICAL TRIAL: NCT00054717
Title: Randomized, Open-label, Comparative Safety and Efficacy Study of Tipranavir Boosted With Low-dose Ritonavir (TPV/RTV) Verses Genotypically-defined Protease Inhibitor/Ritonavir (PI/RTV) in Multiple Antiretroviral Drug-experienced Patients.
Brief Title: Randomized Evaluation of Strategic Intervention in Multidrug Resistant Patients With Tipranavir (RESIST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1182.12
Record Dates: First submitted 2003-02-07; First posted 2003-02-10 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; atazanavir, ritonavir drug combination

ARMS (2):
- Tipranavir(TPV)/low dose ritonavir(r) (Other)
  Interventions: Drug: Tipranavir; Drug: Ritonavir(r)
- Comparator protease inhibitor(CPI)/low dose ritonavir(r) (Other)
  Interventions: Drug: Ritonavir(r); Drug: Comparator Protease Inhibitor (CPI)

INTERVENTIONS:
Drug: Tipranavir
  Arms: Tipranavir(TPV)/low dose ritonavir(r)
Drug: Ritonavir(r)
Drug: Comparator Protease Inhibitor (CPI)
  Arms: Comparator protease inhibitor(CPI)/low dose ritonavir(r)

SUMMARY:
Demonstrate the safety and efficacy of Tipranavir/Ritonavir versus an active treatment regimen in highly treatment experienced Human Immunodeficiency virus 1(HIV-1) infected patients.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be eligible for participation in th is study:

1. Human Immunodeficiency virus 1 (HIV-1) infected males or females >=18 years of age.
2. Screening genotypic resistance report indicating both of the following: at least one primary protease Inhibitor (PI) mutation at the following sites:

30N, 46I/L, 48V, 50V, 82A/F/L/T, 84V or 90M, and no more than two protease mutations on codons 33, 82, 84, or 90.

3. At least 3 consecutive months experience taking antiretrovirals (ARVs) from each of the classes of nucleoside reverse transcriptase inhibitors(NRTI(s)), non-nucleoside reverse transcriptase inhibitors(NNRTI(s)), and protease inhibitors (PIs) at some point in treatment history,with at least 2 protease inhibitor (PI)-based regimens, one of which must be the current regimen, and current protease inhibitor (PI)-based antiretroviral (ARV) medication regimen for at least 3 months prior to randomization.

4. Human Immunodeficiency Virus 1 (HIV-1) viral load >=1,000 copies/mL at screening.

Exclusion criteria:

Patients with any of the following criteria are excluded from participation in t he study:

1. Antiretroviral (ARV) medication naïve.
2. Patients on recent drug holiday, defined as off antiretroviral (ARV) medications for at least 7 consecutive days within the last 3 months.
3. alanine aminotransferase (ALT) >=3.0x upper limit of normal (ULN) and aspartate aminotransferase(AST) >=2.5x upper limit of normal (ULN) (>=Division of AIDS(DAIDS) Grade 1) at either screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2003-01; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (117):
- United States (96):
  - 1182.12.62 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1182.12.108 El Rio SIA, Tucson, Arizona
  - 1182.12.9 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 1182.12.23 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1182.12.12 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 1182.12.76 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1182.12.1 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.12.59 David Geffen School of Medicine at UCLA, Los Angeles, California
  - 1182.12.82 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.12.97 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1182.12.69 UC Davis Medical Center, Sacramento, California
  - 1182.12.89 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1182.12.99 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1182.12.25 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.12.5 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.12.53 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1182.12.98 University of Colorado Health Sciences Center, Denver, Colorado
  - 1182.12.7 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 1182.12.103 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.12.52 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1182.12.70, Washington D.C., District of Columbia
  - 1182.12.79 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1182.12.77 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 1182.12.45 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.12.75 CARES Resource, Miami, Florida
  - 1182.12.85 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1182.12.93 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 1182.12.17 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1182.12.90 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1182.12.63 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.12.78 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1182.12.94 Infectious Disease Research Institute, Tampa, Florida
  - 1182.12.67 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1182.12.123 Infectious Disease Clinics of Emory, Atlanta, Georgia
  - 1182.12.88 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1182.12.72 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1182.12.47 Boehringer Ingelheim Investigational Site, Macon, Georgia
  - 1182.12.8 Family Practice Medical Center, Boise, Idaho
  - 1182.12.105 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.12.3 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.12.49 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1182.12.32 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1182.12.48 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1182.12.33 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1182.12.44 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1182.12.95 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1182.12.81 Boehringer Ingelheim Investigational Site, Portland, Maine
  - 1182.12.30 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1182.12.6 Boehringer Ingelheim Investigational Site, Bethesda, Maryland
  - 1182.12.100 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1182.12.101 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1182.12.41 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1182.12.61 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1182.12.13 University of Michigan Health System, Ann Arbor, Michigan
  - 1182.12.54 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1182.12.56 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1182.12.120 Department of Medicine, HIV/AIDS Program, Minneapolis, Minnesota
  - 1182.12.14 Dybedal Center for Clinical Research, Kansas City, Missouri
  - 1182.12.87 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1182.12.11 Wellness Center, Las Vegas, Nevada
  - 1182.12.4 Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - 1182.12.21 Boehringer Ingelheim Investigational Site, East Orange, New Jersey
  - 1182.12.40 Boehringer Ingelheim Investigational Site, Santa Fe, New Mexico
  - 1182.12.68 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1182.12.34 Boehringer Ingelheim Investigational Site, Mount Vernon, New York
  - 1182.12.119 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.12.22 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.12.36 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.12.58 Beth Israel Medical Center, New York, New York
  - 1182.12.96 Boehringer Ingelheim Investigational Site, New York, New York
  - 1182.12.107 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1182.12.83 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1182.12.43 Boehringer Ingelheim Investigational Site, Valhalla, New York
  - 1182.12.42 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 1182.12.46 Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - 1182.12.109 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1182.12.24 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1182.12.35 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1182.12.65 Ohio State University Medical Center, Columbus, Ohio
  - 1182.12.80 Infectious Disease Institute Clinical Trials Unit, Oklahoma City, Oklahoma
  - 1182.12.114 Pinnacle Health, Harrisburg, Pennsylvania
  - 1182.12.28 University of Pennsylvania, Philadelphia, Pennsylvania
  - 1182.12.50 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1182.12.86 The Miriam Hospital, Providence, Rhode Island
  - 1182.12.10 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1182.12.116 Greenville Hospital System, Greenville, South Carolina
  - 1182.12.2 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1182.12.106 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1182.12.55 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1182.12.31 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1182.12.73 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1182.12.26 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1182.12.91 Boehringer Ingelheim Investigational Site, Annandale, Virginia
  - 1182.12.122 VCU Health Systems, Richmond, Virginia
  - 1182.12.15 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 1182.12.29 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Australia (7):
  - 1182.12.1401 St. Vincent's Hospital, Darlinghurst, New South Wales
  - 1182.12.1405 AIDS Research Initiative / Ground Zero, Darlinghurst, New South Wales
  - 1182.12.1407 Holdsworth House General Practice, Darlinghurst, New South Wales
  - 1182.12.1408 407 Doctors Pty Ltd., Darlinghurst, New South Wales
  - 1182.12.1403 Albion Street Centre, Surry Hills, New South Wales
  - 1182.12.1406 Gold Coast Sexual Health Clinic, Miami, Queensland
  - 1182.12.1404 Alfred Hospital, Melbourne, Victoria
- Canada (13):
  - 1182.12.11002 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1182.12.11010 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1182.12.11016 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1182.12.11012 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1182.12.11001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1182.12.11004 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1182.12.11006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1182.12.11009 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1182.12.11014 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1182.12.11015 Boehringer Ingelheim Investigational Site, Monteal, Quebec
  - 1182.12.11003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1182.12.11007 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1182.12.11013 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- 1182.12.60 Boehringer Ingelheim Investigational Site, Santurce, Puerto Rico

REFERENCES:
- [Derived] Hicks CB, Cahn P, Cooper DA, Walmsley SL, Katlama C, Clotet B, Lazzarin A, Johnson MA, Neubacher D, Mayers D, Valdez H; RESIST investigator group. Durable efficacy of tipranavir-ritonavir in combination with an optimised background regimen of antiretroviral drugs for treatment-experienced HIV-1-infected patients at 48 weeks in the Randomized Evaluation of Strategic Intervention in multi-drug reSistant patients with Tipranavir (RESIST) studies: an analysis of combined data from two randomised open-label trials. Lancet. 2006 Aug 5;368(9534):466-75. doi: 10.1016/S0140-6736(06)69154-X. PMID 16890833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the study there were 630 patients entered as stated in the protocol section. There were 10 patients not treated and are not included within the Participant Flow Module or any other analysis.
Groups:
- Tipranavir(TPV)/Low Dose Ritonavir(r): TPV 500 mg / Ritonavir 200 mg, twice daily
- Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r): lopinavir, amprenavir [or fosamprenavir], saquinavir or indinavir combined with low-dose (100-200 mg) Ritonavir (RTV)
Period: Overall Study
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Started | 313 | 317
Completed | 51 | 18
Not Completed | 262 | 299
Not completed — Randomized but not treated | 2 | 8
Not completed — Adverse Event | 70 | 22
Not completed — Protocol Violation | 18 | 19
Not completed — Lost to Follow-up | 23 | 13
Not completed — Withdrawal by Subject | 32 | 20
Not completed — Other reason not defined above | 117 | 217

BASELINE CHARACTERISTICS:
Population: Safety Set, all patients treated with at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r) | Total
Number analyzed (Participants) | 311 | 309 | 620
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (7.9) | 44.5 (7.1) | 45.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 22 | 55
  Male | 278 | 287 | 565

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response at Week 48
Description: Treatment response (TR) is defined as two consecutive VL ≥ 1 log10 below baseline without discontinuation of study drug, change in anti-retroviral background, or rebound
Time Frame: At week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 33.80 | 16.20
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

2. Primary Outcome: Time to Treatment Failure Through 48 Weeks of Treatment
Description: Time to treatment failure is defined as 0 for patients who never achieve TR otherwise time to treatment failure is the earliest time of death, discontinuation of the study drug or introduction of a new anti-retroviral drug to the regimen if it is not solely related to either toxicity or intolerance clearly attributable to a background, or the first of two consecutive visits with VL measurements <1 log10 below baseline.
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 313 | 317
Days | 113 [0 to 395] | 0 [0 to 171]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

3. Secondary Outcome: Treatment Response at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 41.8 | 23.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

4. Secondary Outcome: Treatment Response at Week 2
Description: as for outcome 1
Time Frame: week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 53.1 | 34.3
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

5. Secondary Outcome: Treatment Response at Week 4
Description: as for outcome 1
Time Frame: week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 52.4 | 33.3
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

6. Secondary Outcome: Treatment Response at Week 8
Description: as for outcome 1
Time Frame: week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 52.4 | 33.3
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

7. Secondary Outcome: Treatment Response at Week 16
Description: as for outcome 1
Time Frame: week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 45.7 | 27.5
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

8. Secondary Outcome: Treatment Response at Week 24
Description: as for outcome 1
Time Frame: week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 42.1 | 23.6
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

9. Secondary Outcome: Treatment Response at Week 32
Description: as for outcome 1
Time Frame: Week 32
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 37.9 | 19.4
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

10. Secondary Outcome: Treatment Response at Week 40
Description: as for outcome 1
Time Frame: Week 40
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 35.4 | 17.8
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

11. Secondary Outcome: Treatment Response at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 33.8 | 16.2
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

12. Secondary Outcome: Treatment Response at Week 56
Description: as for outcome 1
Time Frame: week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 32.5 | 15.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

13. Secondary Outcome: Treatment Response at Week 64
Description: as for outcome 1
Time Frame: week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 31.3 | 15.5
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

14. Secondary Outcome: Treatment Response at Week 72
Description: as for outcome 1
Time Frame: Week 72
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 29.6 | 14.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

15. Secondary Outcome: Treatment Response at Week 80
Description: as for outcome 1
Time Frame: Week 80
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 28 | 14.2
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

16. Secondary Outcome: Treatment Response at Week 88
Description: as for outcome 1
Time Frame: Week 88
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 27.3 | 12.9
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

17. Secondary Outcome: Treatment Response at Week 96
Description: as for outcome 1
Time Frame: Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
percentage of participants | 26.7 | 11.7
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Weighted by the size of enfuvirtide and protease inhibitor strata

18. Secondary Outcome: Time to Treatment Failure Through 96 Weeks of Treatment
Description: as for outcome 2
Time Frame: Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Days | 114 [0 to 858] | 0 [0 to 177]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

19. Secondary Outcome: Time to Confirmed Virologic Failure Through 48 Weeks of Treatment
Description: Time to virologic failure is defined as the time from the start of treatment to the last measurement with a viral load reduction greater than 1.0 log before a confirmed drop of viral load reduction below 1.0 log.
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Days | 113 [0 to 395] | 0 [0 to 174]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

20. Secondary Outcome: Time to Confirmed Virologic Failure Through 96 Weeks of Treatment
Description: as for outcome 19
Time Frame: Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Days | 116 [0 to 858] | 0 [0 to 177]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.0001, Log Rank

21. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Viral Load Nadir, LOCF
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 79.1 | 50.5

22. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 2
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 63.3 | 40.1

23. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 4
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 63.3 | 40.1

24. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 8
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 55.9 | 34.3

25. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 16
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 47.3 | 26.5

26. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 24
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 43.1 | 22.3

27. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 32
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 32
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 38.9 | 19.1

28. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 40
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 40
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 36.7 | 17.5

29. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 48
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 36.3 | 16.2

30. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 56
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 34.1 | 15.5

31. Secondary Outcome: Virologic Response (Viral Load >= 1 Log Drop) at Week 64
Description: Percentage of participants with Viral Load (VL) >= 1 log reduction from baseline
Time Frame: Week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 34.1 | 16.2

32. Secondary Outcome: Median Change From Baseline in Viral Load to Week 2
Time Frame: Baseline to Week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -1.36 [-1.87 to -0.41] | -0.57 [-1.52 to 0]

33. Secondary Outcome: Median Change From Baseline in Viral Load to Week 4
Time Frame: Baseline to Week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -1.56 [-2.15 to -0.45] | -0.46 [-1.71 to 0]

34. Secondary Outcome: Median Change From Baseline in Viral Load to Week 8
Time Frame: Baseline to Week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -1.6 [-2.43 to -0.24] | -0.43 [-1.64 to -0.03]

35. Secondary Outcome: Median Change From Baseline in Viral Load to Week 16
Time Frame: Baseline to Week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -1.08 [-2.5 to -0.18] | -0.32 [-1.26 to -0.03]

36. Secondary Outcome: Median Change From Baseline in Viral Load to Week 24
Time Frame: Baseline to Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.81 [-2.5 to -0.11] | -0.3 [-1.1 to 0.09]

37. Secondary Outcome: Median Change From Baseline in Viral Load to Week 32
Time Frame: Baseline to Week 32
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.73 [-2.42 to -0.06] | -0.24 [-0.87 to 0.09]

38. Secondary Outcome: Median Change From Baseline in Viral Load to Week 40
Time Frame: Baseline to Week 40
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.74 [-2.43 to -0.06] | -0.23 [-0.8 to 0.12]

39. Secondary Outcome: Median Change From Baseline in Viral Load to Week 48
Time Frame: Baseline to Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.61 [-2.34 to -0.04] | -0.24 [-0.81 to 0.12]

40. Secondary Outcome: Median Change From Baseline in Viral Load to Week 56
Time Frame: Baseline to Week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.57 [-2.32 to -0.04] | -0.23 [-0.77 to 0.13]

41. Secondary Outcome: Median Change From Baseline in Viral Load to Week 64
Time Frame: Baseline to Week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.6 [-2.29 to -0.02] | -0.23 [-0.82 to 0.12]

42. Secondary Outcome: Median Change From Baseline in Viral Load to Week 72
Time Frame: Baseline to Week 72
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.65 [-2.29 to -0.05] | -0.21 [-0.76 to 0.12]

43. Secondary Outcome: Median Change From Baseline in Viral Load to Week 80
Time Frame: Baseline to Week 80
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.64 [-2.24 to -0.06] | -0.21 [-0.79 to 0.12]

44. Secondary Outcome: Median Change From Baseline in Viral Load to Week 88
Time Frame: Baseline to Week 88
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.64 [-2.28 to -0.06] | -0.21 [-0.82 to 0.12]

45. Secondary Outcome: Median Change From Baseline in Viral Load to Week 96
Time Frame: Baseline to Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Log(Copies/mL)
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Log(Copies/mL) | -0.6 [-2.24 to -0.01] | -0.21 [-0.76 to 0.13]

46. Secondary Outcome: Mean Change From Baseline to Week 2 in CD4+ Cell Count
Time Frame: Baseline to Week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 23 (48) | 19 (63)

47. Secondary Outcome: Mean Change From Baseline to Week 4 in CD4+ Cell Count
Time Frame: Baseline to Week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 41 (69) | 22 (64)

48. Secondary Outcome: Mean Change From Baseline to Week 8 in CD4+ Cell Count
Time Frame: Baseline to Week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 310 | 309
Cells/mm3 | 49 (72) | 25 (72)

49. Secondary Outcome: Mean Change From Baseline to Week 16 in CD4+ Cell Count
Time Frame: Baseline to Week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 55 (92) | 30 (78)

50. Secondary Outcome: Mean Change From Baseline to Week 24 in CD4+ Cell Count
Time Frame: Baseline to Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 54 (86) | 24 (77)

51. Secondary Outcome: Mean Change From Baseline to Week 32 in CD4+ Cell Count
Time Frame: Baseline to Week 32
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 51 (91) | 26 (87)

52. Secondary Outcome: Mean Change From Baseline to Week 40 in CD4+ Cell Count
Time Frame: Baseline to Week 40
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 50 (100) | 24 (84)

53. Secondary Outcome: Mean Change From Baseline to Week 48 in CD4+ Cell Count
Time Frame: Baseline to Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 46 (95) | 28 (86)

54. Secondary Outcome: Mean Change From Baseline to Week 56 in CD4+ Cell Count
Time Frame: Baseline to Week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 52 (104) | 26 (88)

55. Secondary Outcome: Mean Change From Baseline to Week 64 in CD4+ Cell Count
Time Frame: Baseline to Week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 50 (107) | 26 (94)

56. Secondary Outcome: Mean Change From Baseline to Week 72 in CD4+ Cell Count
Time Frame: Baseline to Week 72
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 50 (113) | 24 (96)

57. Secondary Outcome: Mean Change From Baseline to Week 80 in CD4+ Cell Count
Time Frame: Baseline to Week 80
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 55 (122) | 26 (93)

58. Secondary Outcome: Mean Change From Baseline to Week 88 in CD4+ Cell Count
Time Frame: Baseline to Week 88
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 60 (126) | 29 (100)

59. Secondary Outcome: Mean Change From Baseline to Week 96 in CD4+ Cell Count
Time Frame: Baseline to Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Cells/mm3 | 60 (133) | 28 (97)

60. Secondary Outcome: Time to New CDC Class C Progression Event or Death.
Description: Time to new Centers for Disease Control and Prevention (CDC) class C progression event (i.e., new AIDS defining illness) or death
Time Frame: after 48 weeks of treatment
Population: Safety Analysis Set (SAF), includes all patients treated with at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Days | 448 [448 to 448] | 284 [284 to 284]
Statistical Analysis 1: Comparison: Tipranavir(TPV)/Low Dose Ritonavir(r) vs Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r); Test type: Superiority or Other; p = 0.9894, Log Rank

61. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Viral Load Nadir, LOCF
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 53.4 | 32.4

62. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 2
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 14.8 | 13.6

63. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 4
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 28.3 | 19.1

64. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 8
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 37.3 | 23.6

65. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 16
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 35.7 | 20.7

66. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 24
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 34.4 | 16.5

67. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 32
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: week 32
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 32.8 | 14.9

68. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 40
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 40
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 32.8 | 14.6

69. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 48
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 30.5 | 13.6

70. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 56
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 29.6 | 13.9

71. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 64
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 28.6 | 13.3

72. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 72
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 72
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 28.9 | 12.9

73. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 80
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: Week 80
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 27.7 | 13.6

74. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 88
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: week 88
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 27.7 | 12.6

75. Secondary Outcome: Virologic Response (VL < 400 Copies/ml) at Week 96
Description: Percentage of participants with Viral Load < 400 copies/mL
Time Frame: week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 26.7 | 11.7

76. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Viral Load Nadir, LOCF
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 2 through Week 96 (at any point during trial)
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 37.9 | 20.4

77. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 2
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 2
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 1.9 | 1.9

78. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 4
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 4
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 6.4 | 4.2

79. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 8
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 8
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 16.1 | 8.1

80. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 16
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 16
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 23.5 | 9.4

81. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 24
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 24
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 24.8 | 10

82. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 32
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 32
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 24.8 | 10

83. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 40
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 40
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 23.5 | 8.4

84. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 48
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 48
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 22.5 | 9.7

85. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 56
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 56
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 21.5 | 10

86. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 64
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 64
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 22.8 | 10.7

87. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 72
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 72
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 21.2 | 11.3

88. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 80
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 80
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 20.6 | 10.7

89. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 88
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 88
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 22.2 | 9.7

90. Secondary Outcome: Virologic Response (VL < 50 Copies/ml) at Week 96
Description: Percentage of participants with Viral Load < 50 copies/mL
Time Frame: Week 96
Population: FAS, Full Analysis Set includes all randomized patients treated with at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 311 | 309
Percentage of participants | 20.9 | 9.4

91. Secondary Outcome: Percentage of Patients With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 or 4 Laboratory Abnormalities
Description: NIH Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading Severity of Adult Adverse Experiences, December 2004.
Time Frame: 240 Weeks
Population: Safety Analysis Set with On-Treatment data (SAF-OT), all patients treated with at least one dose of study drug and have on-treatment laboratory values
Measure: Number; unit: Percentage of participants
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Number analyzed (Participants) | 304 | 304
Percentage of participants
  Haemoglobin | 1.3 | 0.7
  White Blood Cell Count Increase | 0 | 0
  White Blood Cell Count Decrease | 5.3 | 5.3
  Platelets | 2.0 | 0.7
  Prothrombin Time | 1.6 | 2.0
  Alanine Transaminase (ALT) | 13.5 | 1.6
  Aspartate Transaminase (AST) | 7.9 | 1.6
  ALT or AST | 15.1 | 2.6
  Bilirubin, Total | 1.0 | 0.7
  Alkaline phosphatase | 1.0 | 0
  Amylase | 11.8 | 9.2
  Lipase | 2.0 | 1.3
  Cholesterol | 23.7 | 8.6
  Triglycerides | 29.3 | 15.5
  Glucose, increase | 3.3 | 2.0
  Glucose, decrease | 0 | 1.0
  Creatinine | 2.0 | 2.3

ADVERSE EVENTS:
Time Frame: up to 240 weeks
Description: Adverse events were monitored throughout the study and reported in the case report form.
Arm/Group | Tipranavir(TPV)/Low Dose Ritonavir(r) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r)
Serious Adverse Events (participants affected / at risk) | 113/311 | 61/309
Other Adverse Events (participants affected / at risk) | 301/311 | 271/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir(TPV)/Low Dose Ritonavir(r) (N=311) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r) (N=309)
Anemia (Blood and lymphatic system disorders) | 6 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Sudden visual loss (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 1
Periproctitis (Gastrointestinal disorders) | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis necrotising (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 4 | 3
Chills (General disorders) | 3 | 0
Cyst (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Granuloma (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Necrosis (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 11 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Immune reconstitution syndrome (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Anogenital warts (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 1
Campylobacter infection (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 2 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 1
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 2 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 2
Disseminated cryptococcosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
End stage AIDS (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 0
Groin abscess (Infections and infestations) | 1 | 0
HIV infection (Infections and infestations) | 3 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 1
Keratitis bacterial (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 3 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 5 | 3
Oral infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 7 | 2
Pneumonia (Infections and infestations) | 13 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Shigella infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 3 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 4 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 1
Drug level increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Volume blood decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 10 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 3 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Convulsion (Nervous system disorders) | 3 | 2
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hemicephalalgia (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Mental retardation (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 3
Drug abuse (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 3
Mental status changes (Psychiatric disorders) | 1 | 0
Fanconi syndrome acquired (Renal and urinary disorders) | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 9 | 2
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1
Vulvar dysplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Drug detoxification (Surgical and medical procedures) | 0 | 1
Intestinal anastomosis (Surgical and medical procedures) | 1 | 0
Intestinal operation (Surgical and medical procedures) | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial rupture (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
Exsanguination (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tipranavir(TPV)/Low Dose Ritonavir(r) (N=311) | Comparitor Protease Inhibitor(CPR)/Low Dose Ritonavir(r) (N=309)
Anaemia (Blood and lymphatic system disorders) | 25 | 6
Abdominal distension (Gastrointestinal disorders) | 27 | 20
Abdominal pain (Gastrointestinal disorders) | 31 | 25
Constipation (Gastrointestinal disorders) | 21 | 13
Diarrhoea (Gastrointestinal disorders) | 123 | 90
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 | 14
Nausea (Gastrointestinal disorders) | 88 | 78
Vomiting (Gastrointestinal disorders) | 56 | 37
Adverse drug reaction (General disorders) | 23 | 19
Fatigue (General disorders) | 71 | 63
Injection site reaction (General disorders) | 30 | 32
Oedema peripheral (General disorders) | 16 | 13
Pain (General disorders) | 19 | 17
Pyrexia (General disorders) | 46 | 27
Bronchitis (Infections and infestations) | 38 | 17
Candidiasis (Infections and infestations) | 16 | 20
Folliculitis (Infections and infestations) | 17 | 10
Influenza (Infections and infestations) | 19 | 5
Nasopharyngitis (Infections and infestations) | 32 | 16
Oral candidiasis (Infections and infestations) | 23 | 13
Sinusitis (Infections and infestations) | 41 | 26
Upper respiratory tract infection (Infections and infestations) | 62 | 37
Urinary tract infection (Infections and infestations) | 16 | 7
Weight decreased (Investigations) | 23 | 21
Decreased appetite (Metabolism and nutrition disorders) | 21 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 29 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 42 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 14
Dizziness (Nervous system disorders) | 27 | 19
Headache (Nervous system disorders) | 53 | 36
Neuropathy peripheral (Nervous system disorders) | 21 | 14
Anxiety (Psychiatric disorders) | 16 | 12
Depression (Psychiatric disorders) | 35 | 26
Insomnia (Psychiatric disorders) | 32 | 30
Erectile dysfunction (Reproductive system and breast disorders) | 16 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 56 | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Night sweats (Skin and subcutaneous tissue disorders) | 18 | 15
Rash (Skin and subcutaneous tissue disorders) | 35 | 33
Hypertension (Vascular disorders) | 16 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.